CLINICAL TRIAL: NCT02097329
Title: A Phase 1, Open-Label, 3-Period Crossover Study Of The Effect Of An Antacid, A Proton Pump Inhibitor And An H2-Receptor Antagonist On Palbociclib (PD-0332991) Bioavailability Under Fed Conditions In Healthy Volunteers
Brief Title: Study Of Three Different Stomach Acid Reducing Agents When Given With Palbociclib (PD-0332991) And Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A5481038
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: bioavailability; antacid; rabeprazole; famotidine; palbociclib
MeSH Terms: interventions — Famotidine; Rabeprazole; Antacids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: Palbociclib under fed conditions (Experimental)
  Interventions: Drug: palbociclib commercial free base; Drug: famotidine; Drug: rabeprazole
- Cohort 2: Palbociclib under fed conditions (Experimental)
  Interventions: Drug: palbociclib commercial free base; Drug: antacid

INTERVENTIONS:
Drug: palbociclib commercial free base — 125 mg oral capsule single dose
  Arms: Cohort 1: Palbociclib under fed conditions
Drug: famotidine — 20 mg oral tablet 10 hours before and 2 hours after palbociclib
  Other Names: Pepcid
  Arms: Cohort 1: Palbociclib under fed conditions
Drug: rabeprazole — 2 x 20 mg oral tablets daily for 6 days then on 7th day, 4 hours after palbociclib
  Other Names: Aciphex
  Arms: Cohort 1: Palbociclib under fed conditions
Drug: palbociclib commercial free base — 125 mg oral capsule single dose
  Arms: Cohort 2: Palbociclib under fed conditions
Drug: antacid — 30 mL orally once (2h before palbociclib)
  Other Names: Mi-Acid Maximum Strength Liquid
  Arms: Cohort 2: Palbociclib under fed conditions
Drug: antacid — 30 mL orally once (2h after palbociclib)
  Other Names: Mi-Acid Maximum Strength Liquid
  Arms: Cohort 2: Palbociclib under fed conditions

SUMMARY:
To investigate the effect of acid reducing agents (an antacid and an H2-receptor antagonist and a proton pump inhibitor) on palbociclib bioavailability in the presence of food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant diseases (hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease).
* Use of tobacco or nicotine containing products within 3 months of screening.
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 6 days
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 6 days

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 6 days
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Apparent Oral Clearance (CL/F) | 6 days
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 6 days
Apparent Volume of Distribution (Vz/F) | 6 days
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Plasma Decay Half-Life (t1/2) | 6 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481038&StudyName=Study%20Of%20Three%20Different%20Stomach%20Acid%20Reducing%20Agents%20When%20Given%20With%20Palbociclib%20%28PD-0332991%29%20And%20Food